CLINICAL TRIAL: NCT05682430
Title: Effects of Speed-based and Mechanical Work Considered HIIT on Physical and Physiological Performance of Chinese Elite Female Referees in Fitness Tests
Brief Title: Speed-based and Mechanical Work Considered HIIT for Football Referees
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Lingling ZHANG, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: ZHANG Lingling
Record Dates: First submitted 2022-11-30; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Physical Fitness
Keywords: high speed interval running; mechanical work

STUDY DESIGN:
Intervention Model Description: In this experiment, the experimental groups conduct the speed-based HIIT with mechanical work. In contrast, the control group take heart rate based HIIT.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heart rate-based HIIT (Active Comparator): 12 weeks heart-rate based HIIT intervention.
  Interventions: Behavioral: Heart rate based HIIT
- VIFT speed-based HIIT with mechanical work (Experimental): 12 weeks VIFT speed-based HIIT with mechanical work.
  Interventions: Behavioral: VIFT speed-based HIIT with mechanical work

INTERVENTIONS:
Behavioral: Heart rate based HIIT — Week1,90% HRmax long duration HIIT + 90% HRmax long duration HIIT. Week2,90% HRmax long duration HIIT + 90% long duration HRmax HIIT. Week3,90% HRmax long duration HIIT + 90% HRmax long duration HIIT. Week4,90% HRmax long duration HIIT + 90% HRmax long duration HIIT. Week5,90% HRmax short duration HIIT + 90～95% HRmax long duration HIIT. Week6,90% HRmax short duration HIIT + 90～95% HRmax long duration HIIT. Week7,90% HRmax short duration HIIT + 90～95% HRmax long duration HIIT. Week8,90% HRmax short duration HIIT + 90～95% HRmax long duration HIIT. Week9,90～95% HRmax short duration HIIT + 90～95% HRmax short duration HIIT. Week10,90～95% HRmax short duration HIIT + 90～95% HRmax short duration HIIT. Week11,90～95% HRmax short duration HIIT + 90～95% HRmax short duration HIIT. Week12,90～95% HRmax short duration HIIT + 90～95% HRmax short duration HIIT.
  Arms: Heart rate-based HIIT
Behavioral: VIFT speed-based HIIT with mechanical work — Week1,Wednesday 65% VIFT HIIT, saturday 65% VIFT HIIT. Week2,Wednesday 65% VIFT HIIT, saturday 65% VIFT HIIT. Week3,Wednesday 67.5% VIFT HIIT, saturday 67.5% VIFT HIIT. Week4,Wednesday 67.5% VIFT HIIT, saturday 67.5% VIFT HIIT. Week5,Wednesday 70% VIFT HIIT, saturday 90% VIFT HIIT. Week6,Wednesday 70% VIFT HIIT, saturday 90% VIFT HIIT. Week7,Wednesday 72.5% VIFT HIIT, saturday 92.5% VIFT HIIT. Week8,Wednesday 72.5% VIFT HIIT, saturday 92.5% VIFT HIIT. Week9,Wednesday 92.5% VIFT HIIT, saturday 100% VIFT HIIT. Week10,Wednesday 92.5% VIFT HIIT, saturday 100% VIFT HIIT. Week11,Wednesday 95% VIFT HIIT, saturday 105% VIFT HIIT. Week12,Wednesday 95% VIFT HIIT, saturday 105% VIFT HIIT.
  Arms: VIFT speed-based HIIT with mechanical work

SUMMARY:
Majority of the existing studies on the high intensity training of referees are heart rate-based prescription. It is probably the most commonly measured physiological marker used to control or measure exercise intensity in the field.Indeed, speed-based intensity training is more acute than heart rate-based training on the intensity of physical work performed above v/pVO2max. This study the setting of exercise intensity reference the ending velocity of the 30-15 intermittent fitness test.

DETAILED DESCRIPTION:
This study was carried out during the 10 weeks of before the seminar which conducted before the season. The assessments were carried out pre and post training intervention in the before and after week of the intervention, it includes 30-15 intermittent fitness test(VIFT),dynamic Yo-Yo intermittent recovery test, 40m repeat speed ability test, change direction test and cooper test.The experimental group(EG) take 10 weeks Speed-based (VIFT) HIIT protocol performed on each Wednesday and Saturday, 60 min for each session. One EG with mechanical work combined in the HIIT exercises, and another EG is not. The control group during the study performed on the same occasion heart rate-based HIIT.

The TL was assessed using the 0-10-point rating perceived exertion (RPE) scale according to the procedures. With the aim to obtain more detailed information especially the muscle strain, during each occasion (i.e., training session or match) the referees should provide differentiated RPE (dRPE) for respiratory (RPEres) and leg muscle (RPEmus) exertion perception.

ELIGIBILITY:
Inclusion Criteria:

* the female referees who register as reserve national degree and above for 2022 and 2023.

Exclusion Criteria:

* Injured
* Any reason can not complete all the required training sessions.

Ages: 23 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-04-22 (Estimated); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
Physical performance in fitness tests | 3 days before the intervention
  Distance covered during dynamic yo-yo test
Physical performance in fitness tests | 3 days before the intervention, just 7min before the dynamic yo-yo test
  The timing consume during the 40m repeat speed ability test
Physical performance in fitness tests | 3 days before the intervention, just 5min before the 40m repeat speed test
  The timing consume during the change of direction test
Physiological performance in the fitness tests | 3days before the intervention
  The HRmax and HRmean and lactic acid concentration during dynamic yo-yo test

SECONDARY OUTCOMES:
Physical performance in fitness tests | 3 days after the 12 weeks intervention
  Distance covered during dynamic yo-yo test, evaluate the participants' ability to repeatedly perform intense exercise.
Physical performance in fitness tests | 3 days after the 12 weeks intervention, 7min before the dynamic yo-yo test
  The timing consume during the 40m repeat speed ability test, evaluate the participants' repeat speed ability.
Physical performance in fitness tests | 3 days after the 12 weeks intervention, 5min before the 40m repeat speed test
  The timing consume during the change of direction test, evaluate the participants' change of direction ability.
Physiological performance in the fitness tests | 3 days after the 12 weeks intervention
  The HRmax and HRmean and lactic acid concentration in dynamic yo-yo test

OTHER OUTCOMES:
Training load | 12 weeks,during each high intensity training
  RPEcr10,RPEmuscle,RPErespiratory
Physical performance in fitness tests | Saturday of the fourth week
  Distance covered during dynamic yo-yo test;The timing consume during the 40m repeat speed ability test;The timing consume during the change of direction test;
Physiological performance in fitness tests | Saturday of the fourth week
  The HRmax and HRmean and lactic acid concentration during dynamic yo-yo test

CONTACTS AND LOCATIONS:
Overall Officials: Lingling ZHANG, Principal Investigator — University Principal Investigator
Locations (1):
- Lingling ZHANG, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No
Since this is my doctoral thesis experiment,I won't share it until I graduate.

REFERENCES:
- [Result] Buchheit M, Laursen PB. High-intensity interval training, solutions to the programming puzzle: Part I: cardiopulmonary emphasis. Sports Med. 2013 May;43(5):313-38. doi: 10.1007/s40279-013-0029-x. PMID 23539308
- [Result] Buchheit M, Laursen PB. High-intensity interval training, solutions to the programming puzzle. Part II: anaerobic energy, neuromuscular load and practical applications. Sports Med. 2013 Oct;43(10):927-54. doi: 10.1007/s40279-013-0066-5. PMID 23832851
- [Result] Billat LV. Interval training for performance: a scientific and empirical practice. Special recommendations for middle- and long-distance running. Part II: anaerobic interval training. Sports Med. 2001 Feb;31(2):75-90. doi: 10.2165/00007256-200131020-00001. PMID 11227980
- [Result] Krustrup P, Bangsbo J. Physiological demands of top-class soccer refereeing in relation to physical capacity: effect of intense intermittent exercise training. J Sports Sci. 2001 Nov;19(11):881-91. doi: 10.1080/026404101753113831. PMID 11695510
- See also: This article is from national library of medicine. — http://pubmed.ncbi.nlm.nih.gov/23539308/
- See also: This article is from national library of medicine. — https://pubmed.ncbi.nlm.nih.gov/23832851/
- See also: This article is from national library of medicine. — https://pubmed.ncbi.nlm.nih.gov/11227980/
- See also: This article is from national library of medicine. — https://pubmed.ncbi.nlm.nih.gov/11695510/